CLINICAL TRIAL: NCT07365059
Title: Clinical Study on Safety and Efficacy of GPRC5D CAR-T Cell Therapy in Relapsed/Refractory Plasma Cell Disorders
Brief Title: Safety and Efficacy of GPRC5D CAR-T Cell Therapy in Relapsed/Refractory Plasma Cell Disorders
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qi deng (Other)
Responsible Party: Sponsor-Investigator, Qi deng, Chief Physician, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XBAP2025-9
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Plasma Cell Dyscrasias
MeSH Terms: conditions — Paraproteinemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPRC5D CAR-T cell intravenous infusion (Experimental)
  Interventions: Biological: GPRC5D CAR-T cell intravenous infusion

INTERVENTIONS:
Biological: GPRC5D CAR-T cell intravenous infusion — GPRC5D CAR-T cell intravenous infusion

SUMMARY:
This study is an open-label, single-arm, dose-escalation and expansion, prospective clinical trial. It enrolls patients with relapsed/refractory plasma cell disorders, administers GPRC5D CAR-T cell therapy, follows up to observe adverse reactions after medication, collects relevant data on treatment efficacy, evaluates the safety and efficacy of CAR-T cells, and simultaneously investigates the cellular kinetic characteristics of CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria：

* According to the World Health Organization (WHO) Classification of Haematopoietic and Lymphoid Tissue Tumours (2022), patients with relapsed/refractory plasma cell disorders that have received adequate treatment and lack effective therapeutic options, including: multiple myeloma, plasma cell leukemia, extramedullary plasmacytoma, solitary plasmacytoma, or primary amyloidosis.i) Relapsed: Disease progression occurs after one or more prior treatments, requiring salvage therapy, and does not meet the criteria for refractory disease.ii) Refractory: No response to initial treatment regimen or salvage therapy, or disease progression within 60 days after treatment. No response is defined as failure to achieve minimal response (MR) or disease progression during treatment.
* The subject's predicted survival time is not less than three months.
* Tumor cells confirmed to be GPRC5D positive by Flow Cytometry (FCM) or Immunohistochemistry.
* The subject failed autologous and allogeneic hematopoietic stem cell transplantation.
* Age 14-75 years (inclusive), both genders eligible.
* ECOG performance status ≤ 2.
* HGB≥70g/L(transfusion permitted).
* The functions of vital organs need to meet the following conditions: ①Creatinine ≤ 2.5 × ULN or Cockcroft-Gault creatinine clearance > 50 ml/min (excluding decreased serum creatinine clearance due to lymphoma mass compression), Combination with hemodialysis treatment is permitted. ②LVEF≥50%,② Oxygen saturation ≥90%,③ SCr≤2.5ULN,④ALT and AST≤3ULN,TBil≤2ULN. In the investigator's judgment, if organ dysfunction is associated with the current disease, the enrollment decision will be made by the investigator.
* Subjects intending to conceive must agree to use contraception prior to study enrollment and for six months post-study. In the event of pregnancy or suspected pregnancy, they should promptly notify the investigator.
* The subject or guardian understands and signs the Informed Consent Form (ICF).

Exclusion Criteria:

Any of the following conditions will not be eligible for enrolment:

* Severe heart failure with left ventricular ejection fraction (LVEF) < 50%.
* History of severe pulmonary function impairment.
* Concurrent other progressive malignant tumors.
* Concurrent severe infection that cannot be effectively controlled.
* Concurrent severe autoimmune disease or congenital immunodeficiency.
* Active hepatitis (hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive with HBV DNA copy number greater than the upper limit of normal at the study center; Anti-HCV positive with HCV-RNA copy number greater than the upper limit of normal at the study center).
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection.
* History of severe allergy to biological products (including antibiotics).
* Received inactivated vaccines such as influenza vaccine, COVID-19 vaccine within 4 weeks prior to screening, or received live attenuated vaccines (such as measles, varicella vaccines) within 8 weeks.
* Allogeneic hematopoietic stem cell transplant patients with persistent acute graft-versus-host disease (GVHD) one month after discontinuation of immunosuppressive agents.
* Patients with other severe physical or mental illnesses or laboratory abnormalities that may increase the risk of study participation or interfere with study results, and patients considered unsuitable for this study by the investigator.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Monitor and record adverse events | up to two years after the CAR-T cell infusion
Overall Response Rate | up to two year after the CAR-T cell infusion

SECONDARY OUTCOMES:
Cell pharmacokinetics Dynamic indicators | up to one month after the CAR-T infusion
  CAR-T/T% by flow cytometry